CLINICAL TRIAL: NCT01868152
Title: Study of Prediction of Opioid Analgesic
Brief Title: The Realtime Detection for Prediction of Opioid Analgesic
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang, Professor, MD., Huazhong University of Science and Technology
Other Study IDs: Predictive opioid
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Surgery; Individuality
Keywords: sufentanil; individual variation; pain threshold; narcotrend index

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aimed to find a quick and timely way to predict the individual variation of efficacy of opioid analgesic during the operation and postoperative analgesia in Chinese patients undergoing elective surgeries. Methods: female patients receiving elective surgery under general anesthesia were recruited into this study. At the time of routine intravenous anesthetic induction we observe the efficacy of opioid analgesic including analgesic effect, effects on Narcotrend index, sedative effect, effects on respiratory system, and aslo effects on cardiovascular system. Then we record the consumption of of opioid analgesic during the operation and postoperative analgesia. Also we record the side effect of the opioid analgesic.

DETAILED DESCRIPTION:
Patients with the following diseases were excluded: known history of chronic pain, psychiatric diseases or communication disorders, diabetes mellitus, severe cardiovascular diseases, kidney or liver diseases with poor hepatic function, alcohol or drug abuse, heavy smoker, pregnancy or at the lactation period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65 years
* Anesthesiologists (ASA) physical status I or II;
* Within ±20% of ideal body weight;
* Agreed to participate the research

Exclusion Criteria: •History of chronic pain;

* Psychiatric diseases;
* Diabetes mellitus;
* Severe cardiovascular diseases;
* Kidney or liver diseases;
* Alcohol or drug abuse (according to the criteria of DSM-IV);
* Pregnancy or at lactation period;
* Disagree to participate to the research

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese female patients receiving elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Rangeability of pressure pain threshold | 8 months
  According to the measurement of pressure pain threshold before and after intravenous injection of opioid analgesics

SECONDARY OUTCOMES:
Rangeability of Narcotrend index | 8 months
  According to the measurement of Narcotrend index before and after intravenous injection of opioid analgesics
Rangeability of Ramsay Sedation Scale | 8 months
  According to the investigation of Ramsay Sedation Scale before and after intravenous injection of opioid analgesics
Rangeability of respiratory frequency | 8 months
  According to the measurement of respiratory frequency before and after intravenous injection of opioid analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xianwei, MD, Study Director — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China